CLINICAL TRIAL: NCT00202228
Title: Lactic Acid Metabolism in HIV-Infected Persons. Predicting Abnormalities in Lactate Production and Clearance Related to Treatment and Liver Disease and Measuring the Impact of Vitamin Supplementation.
Brief Title: Lactate Metabolism Study in HIV Infected Persons
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Ontario HIV Treatment Network (Network)
Responsible Party: Principal Investigator, Dr. Wendy Wobeser, Doctor, Queen's University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DMED-629-02
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: HIV Infections; AIDS; Lactic Acidosis; Lipodystrophy
Keywords: HIV; HIV/AIDS; Lactic Acidosis; Supplementation; Lactate Clearance; Mitochondrial Toxicity; HAART
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Acidosis, Lactic; Lipodystrophy | interventions — Thiamine; Riboflavin; Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Individuals living with HIV who are naive to antiretroviral treatment, or who have been on a treatment interruption for at least six months
  Interventions: Drug: cofactor supplementation (thiamine, riboflavin, L-carnitine)
- 2 (Experimental): Individuals living with HIV who are on an antiretroviral regimen including one of D4T/ddI/ddC/AZT
  Interventions: Drug: cofactor supplementation (thiamine, riboflavin, L-carnitine)
- 3 (Experimental): Individuals living with HIV who are on an antiretroviral regimen including one of D4T/ddI/ddC/AZT and have liver disease.
  Interventions: Drug: cofactor supplementation (thiamine, riboflavin, L-carnitine)
- 4 (Experimental): HIV negative control group
  Interventions: Drug: cofactor supplementation (thiamine, riboflavin, L-carnitine)

INTERVENTIONS:
Drug: cofactor supplementation (thiamine, riboflavin, L-carnitine) — Thiamine: 50 mg po od; Riboflavin: 100 mg po od; L-carnitine: 990 mg po bid.
  Other Names: L-carnitine: Carnitor

SUMMARY:
Lactic acidosis is a potentially life-threatening disease associated with the treatment of chronic HIV infection. Although acidosis is rare, hyperlactatemia is common and may have long term consequences yet to be recognized. Lactic acidosis is a manifestation of mitochondrial toxicity; consequences which have yet to be fully recognized and understood. In this study, we propose to look at lactate clearance and production by two methods, in four treatment groups, including HIV positive subjects on highly active antiretroviral therapy (HAART) treatment regimes and without HAART regimes, with liver steatosis and without, and compared with HIV negative controls. Supplementation with cofactors thiamine, niacin and L-carnitine, which may have a positive effect on lactate metabolism by facilitating mitochondrial function, will be studied as well.

DETAILED DESCRIPTION:
The management of chronic HIV infection is increasingly dependent upon the management of long term toxicities of therapy. Toxicities are often metabolic and include hyperlipidemia, hyperglycemia, osteopenia and lipodystrophy. While more rare, lactic acidosis may present also, and is associated with mortality. The consequences of chronic hyperlactatemia are not well understood, but it is known that the cause is likely related to mitochondrial toxicity of nucleoside analogues, which are the cornerstone class of HIV therapies.

No treatments for the syndrome of chronic lactic acidosis have been proven, but evidence exists which suggests that the utilization of cofactors such as thiamine, riboflavin and L-carnitine in the management of the acute syndrome; these factors may alleviate the mitochondrial compromise.

The mechanism underlying lactic acidemia may be a result of both increased production (as a result of mitochondrial dysfunction), and poor clearance of lactate by the liver which is the primary organ for clearance. Some of this liver dysfunction could also be attributable to mitochondrial toxicity.

In this study we propose to study lactate metabolism among persons with chronic HIV infection (both on treatment and treatment naive) and compare the results to uninfected control population. We will also study a subset of HIV infected persons with known underlying liver disease. Two methodologies will be used: a lactate challenge test and a forearm ischemia test. The effect of supplementation with cofactors which may have a positive effect on lactate metabolism by facilitating mitochondrial function will be studied as well. All persons enrolled for evaluation will have these tests repeated 4-6 weeks after supplementation with standardized doses of cofactors thiamine and L-carnitine between tests. Fat tissue samples and PBMC's will be collected and analyzed for quantity and function, and participants will have liver ultrasounds. Liver biopsies will be completed on those subjects where clinically indicated. The results of the study will provide important insights into the effects on lactate metabolism, nucleoside analogues, and HIV itself.

Our primary hypothesis is that persons on D4T/ddI/ddC/AZT containing highly active antiretroviral therapy (HAART) will demonstrate increased lactate production compared to HIV negative controls; that lactate metabolism will be normalized after treatment with cofactors (riboflavin, thiamine, L-carnitine); that persons with liver disease on therapy will demonstrate prolonged lactate clearance; and that persons changed to a non-D4T/ddI/ddC/AZT containing regime will demonstrate a decrease in lactate production from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Participants at least 18 years of age or older either:

  * HIV negative, or
  * HIV positive, not on antiretroviral therapy (for at least 6 months) or
  * HIV positive, on D4T/ddC/ddI/AZT containing HAART or
  * HIV positive, on D4T/ddC/ddI/AZT containing HAART, with hepatic steatosis/liver disease
* No evidence of acute illness on physical or laboratory examination
* Patients who have voluntarily consented to the study and signed the appropriate consent
* have not been supplementing with multi-vitamins, thiamine, riboflavin for at least 2 months prior to inclusion

Exclusion Criteria:

* Active AIDS defining illness
* Treatment with growth hormone
* Known poor adherence with therapy
* End stage renal disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-07; Primary Completion 2008-10 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Changes in lactate clearance pre and post supplementation | two months

SECONDARY OUTCOMES:
to estimate the change in lactate metabolism and mitochondrial function after a change in antiretroviral therapy to a non D4t/ddC/ddI/AZT regime | six months
Evidence of adverse response to supplements and/or antiretroviral medications | two months (increased where necessary to cover any individual's entire study period should it exceed two months)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wobeser, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada